CLINICAL TRIAL: NCT03282877
Title: Adapting Individual Cognitive Stimulation Therapy (iCST) for Delivery by a Web-application
Brief Title: iCST Web-application for People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iCST web-application
Record Dates: First submitted 2017-07-19; First posted 2017-09-14 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Mild Dementia; Moderate Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCST web-application (Experimental): A computerised cognitive stimulation programme consisting of 21 sessions.
  Interventions: Behavioral: iCST web-application
- Treatment as usual (TAU) (No Intervention): The control group will consist of a treatment-as-usual group and will not receive any additional intervention.

INTERVENTIONS:
Behavioral: iCST web-application — The iCST web-application will be delivered by a carer in regular contact with the person with dementia (family carer, a close friend, or a volunteer befriender) for 1.5 hours a week. It is up to the carer to distribute the time in a matter that is convenient to them (e.g. two long sessions of 45 minutes or 3 shorter sessions of 30 minutes). Participants will be asked to use the web-application for a duration of 11 weeks at their homes. Each session will consist of structured cognitive stimulation aided by the use of multimedia. After completing each session, participants will be guided to a new screen on the web-application in which they will be asked to briefly reflect on the session and provide us with feedback.
  Arms: iCST web-application

SUMMARY:
In the UK, over 670,000 older people are living with dementia which has a substantial, multi-level impact on society, the person with dementia, and their carers. There is a need for an increase in the availability of psychological therapies since people with dementia can face difficulties with staying mentally stimulated and engaged. Cognitive Stimulation Therapy (CST) offers a person based approach and can help to relieve some of these problems. It is a brief manualised evidence based psychological treatment for people with mild to moderate dementia which has shown to improve cognition and quality of life. CST is currently available in both a group and individualised format called iCST. It is worthwhile to explore a computerised version of iCST since it would take together the added value of computer use and the beneficial effects of iCST which might produce combined, positive effects on cognition and quality of life. The investigators have spoken to people with dementia and their carers who are keen on using technology to stay mentally active and stimulated. This study sets out to develop and evaluate the potential benefits of an iCST web-application within a feasibility study. The effects on cognition and quality of life between (a) usual care and (b) iCST web-application over 11 weeks will be compared. A web-application is a website which can easily be accessed on and is compatible with computers and tablets. In order to create the most appropriate and practical web-application, the research team will work closely together with people with dementia, their carers, and the software company. An iCST web-application will compliment traditional CST by making it even more accessible since technology users will be able to access it easily on their device. Furthermore, a computerised version of iCST will by highly relevant for upcoming generations who have grown up with the use of technology.

DETAILED DESCRIPTION:
Scientific justification:

Since the use of technology is rapidly increasing in every aspect of many people's daily lives, previous research has already begun to investigate its application and implementation in multiple areas within dementia care. An example of an area where technology and dementia come together is computerised cognitive interventions. These types of interventions build on the added benefits of computer use such as reduced cognitive decline in older adults and lower risk of receiving a diagnosis of dementia among older men with the added benefits of using one's cognitive capacities. In a recent systematic review, Garcia-Casal et al. (2016) concluded that computerised cognitive interventions led to significant improvements in cognition, depression and anxiety among people with dementia. Computerised cognitive interventions may have more of an impact on cognition than non-computerised cognitive interventions.

In a randomised pilot trial conducted by Tárraga et al. (2006) which was included in Garcia-Casal's review, people with mild Alzheimer's Disease were allocated to a treatment group and a control group. The treatment group consisted of both a computerised cognitive stimulation programme and a non-computerised, face-to-face cognitive stimulation programme delivered in groups. The control group consisted solely of the non-computerised, cognitive stimulation programme. The results showed that that people with mild Alzheimer's Disease showed greater improvements in cognition lasting for 24 weeks in the treatment group which suggests added benefits of a computerised cognitive stimulation programme.

These positive findings suggest that it is worthwhile to continue conducting research in the area of computerised cognitive interventions. Interestingly, Garcia-Casal et al (2016) have pointed out that the area of computerised cognitive stimulation (which is an area of computerised cognitive interventions) is relatively underdeveloped. Most computerised cognitive interventions are geared towards cognitive training.

At the moment there are multiple, paper-based cognitive stimulation interventions available of which Cognitive Stimulation Therapy is being used more predominantly in the UK. CST is a brief evidence-based psychological treatment for people with mild to moderate dementia. It consists of mentally stimulating and engaging group activities which have shown to improve cognition and quality of life in a large scale randomised controlled trial. More recently, an individualised version of CST (iCST) was developed which is a home-based version of CST administered by informal carers (e.g., friends, family members). The content of the sessions is similar to those of CST. A multi-centre RCT of iCST showed no improvements in cognition and QoL for people with dementia, nor evidence of improvements in carers' mental and physical health. However, people with dementia receiving iCST reported a better relationship quality with their carer, and carers reported an improved health-related QoL. These findings indicate a need for further research to determine the effectiveness of carer-led cognitive stimulation interventions for people with dementia since most people received fewer than recommended number of iCST due to low adherence.

Since there is a need for more research in both the area of computerised cognitive stimulation and carer-led cognitive stimulation, this research sets out to develop and evaluate the potential benefits of iCST adapted for delivery by an interactive (touch-screen) web-application in a feasibility study. The investigators are setting out to combine the added value of computer use and the beneficial effects of CST/iCST in order to produce benefits in cognition and quality of life. A participatory process while developing the web-application in the form of consultations, focus groups and interviews will be employed. Preliminary consultations with people with dementia and their carers have already given the investigators information on attitudes towards (touch-screen) technology, both appealing and non-appealing features of applications and desired length/duration of iCST.

The investigators hope to see signs of improvements in quality of life and cognition after using the iCST web-application. If this is the case, this could lead to a larger randomised controlled trial with more participants to formally establish effectiveness. An iCST web-application has the potential to be more accessible for people on a national and an international level when adapted to appropriate cultural contexts compared to paper-based manuals. Lastly, the iCST web-application could be used long-term and could rapidly become widely used as a clinically and cost-effective standardised, and feasible intervention.

Design and methodology:

1. The focus groups and interviews will be a multi-centre study to gain insights and perspectives from people with dementia and their carers regarding the usability of the iCST web-app. This will enable the investigators to optimise the developmental process and learn about the experiences of the participants while they interact with the web-application. Observational and transcribed audio-recorded data will be collected from the focus groups and interviews which will be semi-structured in nature.
2. The feasibility study will be a multicentre, pragmatic, single blind, randomised 2 treatment arm (iCST web-app vs treatment as usual) study over 11 weeks.

In accordance with good research practice, the investigators have decided to run a feasibility study prior to running a larger randomised controlled trial in order to assess the usability of the iCST web-application and the feasibility of running a larger-scale randomised clinical trial. With this feasibility study the investigators will be able to gain insights with regard to recruitment/drop-out rates, adherence, sample size, appropriateness of outcome measures, changes to made to the web-application etc. This will all be necessary information before a larger trial can be conducted.

Programme development:

The iCST web-application will be adapted from the paper-based iCST manual. The amount of sessions will be reduced from 75 to 21 after consultations with people with dementia and carers pointed out that the paper-based iCST manual contained too many sessions. Multimedia within the web-application will be used and participants will be given the opportunity to provide ongoing feedback on the web-application itself after completing each session. The research team will work together with all the stakeholders such as the software company employed to build the web-application, the people with dementia, and their carers. Regular consultations, focus groups and interviews should aid the development of the web-application in ensuring it is feasible, practical and appealing.

Recruitment for the study:

Recruitment for the focus groups, interviews and feasibility study will take place in a variety of community settings in Nottingham consisting of both primary care settings (outpatient clinics) and secondary care settings (community mental health teams (CMHTs), memory clinics, care homes, day centres, and voluntary sector organizations such as the Alzheimer's Society). By including a variety of settings, the reach for people with dementia and their carers will be extended. The PhD student will make close links with the aforementioned services and organisations through attendance and regular contact. In addition, the distribution of information leaflets and posters to organisations and professionals involved in the identification of possible participants will facilitate the recruitment process.

The initial approach will be from a member of the person with dementia's usual care team. If the person with dementia and carer are willing and suitable for participation, the PhD student will fully inform them about of all aspects pertaining to involvement in the study through in person conversations and information leaflets. It will be explained to the potential participant that; (i) entry into the study is entirely voluntary and that their treatment and care will not be affected by their decision, (ii) they can withdraw at any time but attempts will be made to avoid this occurrence and (iii) in the event of their withdrawal their data collected so far cannot be erased and we will seek consent to use the data in the final analyses where appropriate.

Sample size:

The sample size estimation for the focus groups and interviews is based on previous work in the iCST study. For the current study, four focus groups with six participants each (one with people with dementia, one with carers, two collaborative groups) and ten interviews (five with people with dementia and five with carers) will be conducted.

The investigators have estimated the sample size to be 60 participants. This is partly based on previous work with iCST considering the numbers recruited and the amount of centres involved in the iCST trial. The iCST trial recruited 356 participants over eight sites across the UK (Bangor, Devon, Dorset, Hull, Lincolnshire, London, Manchester, Norfolk and Suffolk). This equals to an average of 45 dyads per site. We will have an equal distribution of dyads across the two groups leading to 30 dyads per arm (iCST web-application vs. treatment-as-usual). The field-testing phase of iCST (without a control group) included 22 dyads which roughly resembles the sample size for the current feasibility study.

A sample size of 60 participants will be sufficient to demonstrate the effectiveness of the iCST web-application with an effect size of 0.80 with 80% power and 5% significance (two-tailed). The effect size has been chosen based on the sample size.

Timetable:

Focus groups/interviews (start from May 2018 onwards):

1. 3 months recruitment;
2. 4 months running of groups and interviews in Nottingham recruitment
3. 6 months analysis and writing up findings

Feasibility trial (start from November 2018 onwards):

1. 5 months of recruitment;
2. 7 months of running feasibility study;
3. 5 months analysis and writing up findings

ELIGIBILITY:
Inclusion Criteria:

Person with dementia:

* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria for dementia (American Psychiatric Association, 2013).
* Score 10 or above on the Mini Mental State Examination (MMSE) (Folstein, Folstein, & McHugh, 1975) or score of 16 or above on the Montreal Cognitive Assessment (MoCA) (Trzepacz et al., 2015) where available.
* Some ability to communicate and understand (e.g. ability to give informed consent)
* Ability to speak and understand English
* See/hear well enough to participate
* No major physical illness or disability affecting their participation
* Age range: 50 years - no maximum age limit
* Availability of a tablet to the person with dementia and carer
* Availability of a carer (or friend/befriender) to participate in the focus groups, interviews and iCST web-app sessions

Carer:

* Minimum age: 21
* Ability to speak and understand English
* See/hear well enough to participate
* No major physical illness or disability affecting their participation

Exclusion criteria

Person with dementia and carer:

- Concurrent participation in any other interventional study for people with dementia/carers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cognition (person with dementia) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  ADAS-Cog: to measure the severity of the cognitive symptoms (memory, language, praxis, attention and other cognitive abilities)
Change in quality of life (person with dementia) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  QoL-AD: self reporting questionnaire to investigate: physical health, energy, mood, living situation, memory, marriage, friends, chores, fun, money, self and life).
Change in general health outcome (carer) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  EQ-5D: An instrument used to measure health outcome, it provides a descriptive profile for health status. It evaluates quality of life in carers.

SECONDARY OUTCOMES:
Depression (person with dementia) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  CSDD: to measure depressive symptoms: mood-related signs, behavioural disturbances, physical signs, biological functions and ideational disturbances
Behavioural symptoms (person with dementia) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  NPI: to asses 10 behavioural disturbances: delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy and aberrant motor activity.
Activities of daily living (person with dementia) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  BADLS: BADLS is an instrument consisting of 20 daily-living abilities (basic and instrumental activities)
Relation between person with dementia and carer (both) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  QPCR: a measure of relationship quality which will be completed by both the person with dementia and the carer
Depression/anxiety (carer) | Pre-intervention (baseline), 5 weeks post baseline, 11 weeks post baseline
  HADS: is a useful measure anxiety and depression for carer. It consists of 14 questions (7 for anxiety and 7 for depression).

OTHER OUTCOMES:
Computer use self efficacy | Pre-intervention (baseline)
  CUSE: will be used to assess self-efficacy beliefs in the context of computer/tablet use
System usability | 11 weeks post baseline
  SUS: is a widely-used questionnaire measuring the usability of a technology-based tool e.g. a computer program or other device.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Orrell, MD, PhD, Study Chair — University of Nottingham; Justine Schneider, PhD, Study Director — University of Nottingham; Harleen Rai, MSc., Principal Investigator — University of Nottingham; Lauren Yates, PhD, Study Director — University of Nottingham
Locations (4):
- United Kingdom (4):
  - Derbyshire Healthcare NHS Foundation Trust, Derby, Derbyshire
  - Leicestershire Partnership NHS Trust, Leicester, Leicestershire
  - Lincolnshire Partnership NHS Foundation Trust, Lincoln, Lincolnshire
  - Nottinghamshire Healthcare NHS Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xavier AJ, d'Orsi E, de Oliveira CM, Orrell M, Demakakos P, Biddulph JP, Marmot MG. English Longitudinal Study of Aging: can Internet/E-mail use reduce cognitive decline? J Gerontol A Biol Sci Med Sci. 2014 Sep;69(9):1117-21. doi: 10.1093/gerona/glu105. PMID 25116923
- [Background] Almeida OP, Yeap BB, Alfonso H, Hankey GJ, Flicker L, Norman PE. Older men who use computers have lower risk of dementia. PLoS One. 2012;7(8):e44239. doi: 10.1371/journal.pone.0044239. Epub 2012 Aug 28. PMID 22937167
- [Background] Garcia-Casal JA, Loizeau A, Csipke E, Franco-Martin M, Perea-Bartolome MV, Orrell M. Computer-based cognitive interventions for people living with dementia: a systematic literature review and meta-analysis. Aging Ment Health. 2017 May;21(5):454-467. doi: 10.1080/13607863.2015.1132677. Epub 2016 Jan 25. PMID 26806365
- [Background] Tarraga L, Boada M, Modinos G, Espinosa A, Diego S, Morera A, Guitart M, Balcells J, Lopez OL, Becker JT. A randomised pilot study to assess the efficacy of an interactive, multimedia tool of cognitive stimulation in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2006 Oct;77(10):1116-21. doi: 10.1136/jnnp.2005.086074. Epub 2006 Jul 4. PMID 16820420
- [Background] Hodge, S., Hailey, E & Orrell, M. (eds) (2014). Memory Services National Accreditation Programme - Standards for Memory Services (4th Edition). London: Royal College of Psychiatrists.
- [Background] Spector, A., Thorgrimsen, L., Woods, B., & Orrell, M. (2006). Making a difference. London: Hawker Publications.
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Orrell M, Yates L, Leung P, Kang S, Hoare Z, Whitaker C, Burns A, Knapp M, Leroi I, Moniz-Cook E, Pearson S, Simpson S, Spector A, Roberts S, Russell I, de Waal H, Woods RT, Orgeta V. The impact of individual Cognitive Stimulation Therapy (iCST) on cognition, quality of life, caregiver health, and family relationships in dementia: A randomised controlled trial. PLoS Med. 2017 Mar 28;14(3):e1002269. doi: 10.1371/journal.pmed.1002269. eCollection 2017 Mar. PMID 28350796
- [Background] Yates LA, Orrell M, Spector A, Orgeta V. Service users' involvement in the development of individual Cognitive Stimulation Therapy (iCST) for dementia: a qualitative study. BMC Geriatr. 2015 Feb 6;15:4. doi: 10.1186/s12877-015-0004-5. PMID 25655940
- [Background] Orrell M, Aguirre E, Spector A, Hoare Z, Woods RT, Streater A, Donovan H, Hoe J, Knapp M, Whitaker C, Russell I. Maintenance cognitive stimulation therapy for dementia: single-blind, multicentre, pragmatic randomised controlled trial. Br J Psychiatry. 2014 Jun;204(6):454-61. doi: 10.1192/bjp.bp.113.137414. Epub 2014 Mar 27. PMID 24676963
- [Background] Yates LA, Leung P, Orgeta V, Spector A, Orrell M. The development of individual cognitive stimulation therapy (iCST) for dementia. Clin Interv Aging. 2014 Dec 30;10:95-104. doi: 10.2147/CIA.S73844. eCollection 2015. PMID 25565792
- [Derived] Rai HK, Schneider J, Orrell M. An Individual Cognitive Stimulation Therapy App for People with Dementia and Carers: Results from a Feasibility Randomized Controlled Trial (RCT). Clin Interv Aging. 2021 Dec 22;16:2079-2094. doi: 10.2147/CIA.S323994. eCollection 2021. PMID 35221680
- [Derived] Rai HK, Schneider J, Orrell M. An Individual Cognitive Stimulation Therapy App for People With Dementia and Their Carers: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2021 Apr 8;10(4):e24628. doi: 10.2196/24628. PMID 33830058